CLINICAL TRIAL: NCT03893955
Title: A Phase 1, Multicenter, Open-Label Study to Determine the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Combinations of ABBV-927 With ABBV-368, Budigalimab (ABBV-181) and/or Chemotherapy in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Determine the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ABBV-927 With ABBV-368, Budigalimab (ABBV-181) and/or Chemotherapy in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M19-037; 2019-000478-45 (EudraCT Number)
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Advanced Solid Tumors; Triple-Negative Breast Cancer (TNBC); Non-small-cell-lung-cancer (NSCLC); Metastatic Solid Tumors
Keywords: Cancer; Advanced Solid Tumors; Triple-Negative Breast Cancer (TNBC); Non-small-cell-lung-cancer (NSCLC); ABBV-927; ABBV-368; ABBV-181; metastatic solid tumors; dose-escalation; recommended phase 2 dose; budigalimab
MeSH Terms: conditions — Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — budigalimab; Carboplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Dose Escalation Arm A: ABBV-927 + ABBV-368 Solid Tumors (Experimental): Participants with Solid Tumors will receive various doses of ABBV-927 by intravenous (IV) infusion plus ABBV-368. This will determine the recommended phase two dose (RP2D) of ABBV-927.
  Interventions: Drug: ABBV-927; Drug: ABBV-368
- Dose Escalation Arm B: ABBV-927 + ABBV-368 + ABBV-181 NSCLC (Experimental): Participants with non-small-cell-lung-cancer (NSCLC) will receive ABBV-927 IV at various dose levels + ABBV-368 + ABBV-181. This will determine the recommended phase two dose (RP2D) of ABBV-927 + ABBV-368 + ABBV-181.
  Interventions: Drug: ABBV-927; Drug: ABBV-368; Drug: ABBV-181
- Dose Expansion Arm 1: ABBV-927 + Carboplatin + ABBV-368 TNBC (Experimental): Participants with Triple Negative Breast Cancer (TNBC) will receive ABBV-927 (at the RP2D established in Arm A) + Carboplatin + ABBV-368 by IV.
  Interventions: Drug: ABBV-927; Drug: ABBV-368; Drug: Carboplatin
- Dose Expansion Arm 2: ABBV-927 + Carboplatin + ABBV-181 TNBC (Experimental): Participants with TNBC will receive ABBV-927 (at the RP2D established in Arm A) + Carboplatin + ABBV-181 by IV.
  Interventions: Drug: ABBV-927; Drug: ABBV-181; Drug: Carboplatin
- Dose Expansion Arm 3: ABBV-927 + Carboplatin TNBC (Experimental): Participants with TNBC will receive ABBV-927 (at the RP2D established in Arm A) + Carboplatin by IV.
  Interventions: Drug: ABBV-927; Drug: Carboplatin
- Dose Expansion Arm 4: ABBV-927+ Nab-paclitaxel + ABBV-368 TNBC (Experimental): Participants with TNBC will receive ABBV-927 (at the RP2D established in Arm A) + Nab-paclitaxel + ABBV-368 by IV.
  Interventions: Drug: ABBV-927; Drug: ABBV-368; Drug: Nab-paclitaxel
- Dose Expansion Arm 5: ABBV-927 + ABBV-368 + ABBV-181 NSCLC (Experimental): Participants with NSCLC will receive ABBV-927 (at the RP2D established in Arm B) + ABBV-368 + ABBV-181 by IV.
  Interventions: Drug: ABBV-927; Drug: ABBV-368; Drug: ABBV-181

INTERVENTIONS:
Drug: ABBV-927 — Intravenous (IV) Infusion
Drug: ABBV-368 — Intravenous (IV) Infusion
  Arms: Dose Escalation Arm A: ABBV-927 + ABBV-368 Solid Tumors; Dose Escalation Arm B: ABBV-927 + ABBV-368 + ABBV-181 NSCLC; Dose Expansion Arm 1: ABBV-927 + Carboplatin + ABBV-368 TNBC; Dose Expansion Arm 4: ABBV-927+ Nab-paclitaxel + ABBV-368 TNBC; Dose Expansion Arm 5: ABBV-927 + ABBV-368 + ABBV-181 NSCLC
Drug: ABBV-181 — Intravenous (IV) Infusion
  Other Names: Budigalimab
  Arms: Dose Escalation Arm B: ABBV-927 + ABBV-368 + ABBV-181 NSCLC; Dose Expansion Arm 2: ABBV-927 + Carboplatin + ABBV-181 TNBC; Dose Expansion Arm 5: ABBV-927 + ABBV-368 + ABBV-181 NSCLC
Drug: Carboplatin — Intravenous (IV) Infusion
  Arms: Dose Expansion Arm 1: ABBV-927 + Carboplatin + ABBV-368 TNBC; Dose Expansion Arm 2: ABBV-927 + Carboplatin + ABBV-181 TNBC; Dose Expansion Arm 3: ABBV-927 + Carboplatin TNBC
Drug: Nab-paclitaxel — Intravenous (IV) Infusion
  Arms: Dose Expansion Arm 4: ABBV-927+ Nab-paclitaxel + ABBV-368 TNBC

SUMMARY:
A study evaluating the safety, pharmacokinetics (PK), pharmacodynamics, and preliminary efficacy of ABBV-927 with ABBV-368, Budigalimab (ABBV-181) and/or chemotherapy in participants with selected solid tumors. This study consists of 2 main parts, a dose-escalation phase and a dose-expansion phase. The dose-expansion phase can begin once the recommended phase 2 dose/maximum tolerated dose (RP2D/MTD) is determined in the dose-escalation phase.

ELIGIBILITY:
Inclusion Criteria:

* Adequate liver, kidney and hematology function as demonstrated by laboratory values detailed in the study protocol.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Dose-Escalation:

* Arm A: Participants with an advanced solid tumor who have progressed on standard therapies known to provide clinical benefit and/or participants who have refused or are intolerant of such therapy.
* Arm B (non-small-cell-lung-cancer [NSCLC]): Participants with histologically or cytologically confirmed NSCLC who previously progressed during or after an anti-programmed cell death (PD)-1 or PD ligand 1 (PD-L1) therapy and a platinum-based regimen in the recurrent or metastatic setting.

Dose-Expansion:

* Arm 1, 2, and 3 (triple-negative breast cancer [TNBC]): Participants with histologically or cytologically confirmed breast adenocarcinoma that is estrogen receptor/progesterone receptor/human epidermal growth factor receptor (HER)2-negative who must have disease progression during or after at least 1 systemic therapy that included a taxane in the metastatic or recurrent setting and who are treatment-naïve to immunotherapy.
* Arm 4 (TNBC): Participants with histologically or cytologically confirmed TNBC who have received no previous anti-cancer therapy for TNBC, and who are PD-L1 negative on tumor tissue by immunohistochemistry (IHC) assay.
* Arm 5 (NSCLC): Participants with histologically or cytologically confirmed NSCLC who previously progressed either during or after an anti-PD-1 or PD-L1 therapy and a platinum-based regimen in the recurrent or metastatic setting.

Exclusion Criteria:

* Has history of inflammatory bowel disease or pneumonitis.
* Has uncontrolled metastases to the central nervous system.
* Has a concurrent malignancy that is clinically significant, treatment is required, or the participant is not clinically stable.
* Has had a major surgery ≤ 28 days prior to the first dose of study drug or the surgical wound is not fully healed.
* Has previously treated with an anti-PD- or PD-L1-targeting agent and had during the course of their therapy:
* any immune-mediated toxicity of Grade 3 or worse severity
* treatment of the toxicity with systemic corticosteroids
* any hypersensitivity to the PD-1 or PD-L1-targeting agent
* any treatment-related toxicity resulting in discontinuation of the PD-1 or PD-L1 targeting agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Dose Expansion: Objective Response Rate (ORR) | Up to approximately 2 years following the first dose of study drug
  ORR is defined as the percentage of participants with either complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Dose-Escalation Phase: Recommended Phase 2 Dose (RP2D) of ABBV-927 + ABBV-368 | Up to approximately 6 months
  The RP2D of ABBV-927 + ABBV-368 will be determined during the dose-escalation phase of the study. RP2D will be determined using available safety and pharmacokinetics data.
Dose-Escalation Phase: Recommended Phase 2 Dose (RP2D) of ABBV-927 + ABBV-368 + ABBV-181 | Up to approximately 6 months
  The RP2D of ABBV-927 + ABBV-368 + ABBV-181 will be determined during the dose-escalation phase of the study. RP2D will be determined using available safety and pharmacokinetics data.

SECONDARY OUTCOMES:
Dose-Expansion Phase: Progression-free Survival (PFS) | Up to approximately 2 years since the first dose of study drug
  PFS is defined as the time from date of first study drug exposure to disease progression or death, whichever occurs first.
Dose-Expansion Phase: Duration of Response (DOR) | Up to approximately 2 years since the first dose of study drug
  DOR defined as the time from the participant's initial response to study drug therapy to disease progression or death, whichever occurs first.
Maximum Serum Concentration (Cmax) | Up to approximately 12 weeks after participant's initial dose of study drug
  Maximum Serum Concentration (Cmax)
Time to Maximum Observed Serum Concentration (Tmax) | Up to approximately 12 weeks after participant's initial dose of study drug
  Time to Maximum Observed Serum Concentration (Tmax)
Area Under the Serum Concentration Versus Time Curve from Time 0 to the Time of the Last Measurable Concentration (AUCτ) | Up to approximately 12 weeks after participant's initial dose of study drug
  Area under the serum concentration versus time curve from time 0 to the time of the last measurable concentration (AUCτ).
Terminal Phase Elimination Half-life (t1/2) | Up to approximately 4 weeks after participant's initial dose of study drug
  Terminal Phase Elimination Half-life (t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (26):
- United States (13):
  - Highlands Oncology Group, PA /ID# 218863, Springdale, Arkansas
  - St Jude Hospital dba St Joseph /ID# 211130, Santa Rosa, California
  - Yale University School of Medicine /ID# 210678, New Haven, Connecticut
  - Moffitt Cancer Center /ID# 215037, Tampa, Florida
  - Fort Wayne Medical Oncology and Hematology, Inc /ID# 226072, Fort Wayne, Indiana
  - Washington University-School of Medicine /ID# 221399, St Louis, Missouri
  - Duke Cancer Center /ID# 217641, Durham, North Carolina
  - Carolina BioOncology Institute /ID# 210664, Huntersville, North Carolina
  - UPMC Hillman Cancer Ctr /ID# 222747, Pittsburgh, Pennsylvania
  - Tennessee Oncology-Nashville Centennial /ID# 221400, Nashville, Tennessee
  - Mary Crowley Cancer Research /ID# 210716, Dallas, Texas
  - NEXT Oncology /ID# 210717, San Antonio, Texas
  - Virginia Cancer Specialists - Fairfax /ID# 210671, Fairfax, Virginia
- Duplicate_Icon Cancer Centre /ID# 224084, South Brisbane, Queensland, Australia
- France (5):
  - Institut de Cancérologie de l'Ouest René Gauducheau /ID# 212880, Saint-Herblain, Loire-Atlantique
  - Institut Curie /ID# 223475, Paris, Paris
  - Centre Leon Berard /ID# 217910, Lyon, Rhone
  - Centre Jean Perrin /ID# 217911, Clermont-Ferrand
  - AP-HP - Hopital Bichat - Claude-Bernard /ID# 212869, Paris
- The Chaim Sheba Medical Center /ID# 211699, Ramat Gan, Tel Aviv, Israel
- Spain (4):
  - Hospital Universitario Vall d'Hebron /ID# 212804, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 212806, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 212805, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 221671, Málaga
- Taiwan (2):
  - National Taiwan University Hospital /ID# 210993, Taipei City, Taipei
  - China Medical University Hospital /ID# 221090, Taichung

IPD SHARING:
Plan to Share IPD: No